CLINICAL TRIAL: NCT02448992
Title: Neuropsychological and Oncological Outcomes After Hippocampal-Sparing Prophylactic Cranial Irradiation in Postoperative Patients With Pathologically Nodal Positive Non-Small-Cell Lung Cancer - A Prospective Follow-up Study
Brief Title: Hippocampal-Sparing Prophylactic Cranial Irradiation in Pathologically Nodal Positive Non-Small-Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103-6591A3
Record Dates: First submitted 2015-04-13; First posted 2015-05-20 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Non-Small-Cell Lung Cancer (NSCLC); Brain Metastasis
Keywords: Neurobehavioral Assessments; Neurocognitive Functions (NCF); Prophylactic Cranial Irradiation (PCI); Hippocampus; Hippocampal-Sparing PCI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

ARMS (2):
- PCI via hippocampal-sparing WBRT (Experimental): All studied patients should undergo a computed tomography (CT) simulation scan encompassing the entire head region with 1.25-mm slice thickness using a thermoplastic mask for immobilization. To achieve conformal hippocampal sparing during the delivery of WBRT, the technique of volumetric modulated arc therapy (VMAT) via Linac-based RapidArc® or TrueBeamTM is employed in our treatment planning. All treatment plans are delivered by using the Linac Varian-iX or TrueBeamTM. In terms of dose prescription, a dose of 30 Gy in 15 fractions is prescribed to whole-brain planning target volume (PTV) under the setting of prophylactic cranial irradiation for NSCLC patients.
  Interventions: Radiation: hippocampal-sparing WBRT
- observation without PCI (No Intervention)

INTERVENTIONS:
Radiation: hippocampal-sparing WBRT
  Arms: PCI via hippocampal-sparing WBRT

SUMMARY:
Background. During the clinical course of patients with locoregionally advanced non-small-cell lung cancer (LA-NSCLC) who have undergone aggressive treatment, brain metastasis (BM) is a frequent seen pattern of disease relapse, which cannot be ignored. It still remains unresolved whether prophylactic cranial irradiation (PCI) via whole brain radiotherapy (WBRT) should be recommended for NSCLC patients with stage III or pathologically nodal positive disease. Actually, PCI would significantly decrease the incidence of BM; however, potential WBRT-related neurocognitive function (NCF) sequelae are indeed a concern, which has made PCI seldom applied in clinical practice. In terms of the time course of WBRT-induced NCF decline, it might vary considerably according to the specific domains which are selected to be measured. Early neurocognitive decline principally involve impairments of episodic memory, which has been significantly associated with functions of the hippocampus. This study thus aims to explore the impact of PCI on the subsequent risk of developing BM and the multi-domain neurobehavioral functions in our eligible patients.

Methods. Potentially eligible subjects are postoperative NSCLC patients with a status of pathologically nodal metastasis (pN+). Patients randomly assigned to the PCI arm will undergo the course of hippocampal-sparing PCI after they complete the fourth course of adjuvant platinum-based chemotherapy. Radiotherapy dose will be 3000 cGy in 15 fractions during three weeks. Except for the administration of hippocampal-sparing PCI, patients assigned to the observation arm should receive the same baseline and follow-up brain imaging examinations and neurocognitive assessments as those in PCI arm. Accordingly, a battery of neuropsychological measures, which includes 7 standardized neuropsychological tests (e.g., executive functions, verbal & non-verbal memory, working memory, and psychomotor speed), is used to evaluate neurobehavioral functions for our registered patients.

Expected results. This randomized controlled study aims to verify that the incidence of BM still can significantly be reduced by hippocampal-sparing PCI; additionally, NCF preservation regarding neurobehavioral assessments might also be achieved by hippocampal-sparing PCI as compared with the observation arm without PCI. No matter what the final results present, it is believed that this randomized controlled trial (RCT) will provide us solid evidence concerning the exact value of hippocampal-sparing PCI in our patient setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NSCLC
* Must be adult patients (≥ 18 years old) who have received definitive surgery and have a permanent pathology of nodal metastasis
* Platinum-based chemotherapy is mandatory
* Good performance status better than Eastern Cooperative Group (ECOG) of 2 or a general status of Karnofsky (KPS) > 70 %
* Should have sufficient proficiency in Mandarin language

Exclusion Criteria:

* Have received prior cranial irradiation
* Presence of other active primary cancer (exception of basal cell carcinoma of skin and cervical carcinoma in situ)
* Radiographic evidence of brain metastasis/metastases
* Clinical evidence of extracranial metastatic disease
* Hypersensitivity to magnetic resonance (MR) contrast enhancer
* Serious medical or psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
time to the development of brain metastasis/metastases (BM), irrespective of the absence of active neurological symptoms | one year

SECONDARY OUTCOMES:
the effects of hippocampal-sparing PCI on neurocognitive functions (NCF) | up to 18 months
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in either verbal memory [Wechsler Memory Scale - 3rd edition (WMS III) - Word List score] or non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of the course of WBRT with hippocampus avoidance (HA-WBRT). Additionally, the follow-up of neurocognitive assessment will also be administered at 12 months and up to 18 months after the start of PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Cheng Yang, Ph.D., Principal Investigator — Chang Gung University; Shinn-Yn Lin, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan